CLINICAL TRIAL: NCT07315334
Title: Assessing Functional Impairments in Patients With Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Brief Title: Assessing Functional Impairments in Patients With Chemotherapy-Induced Peripheral Neuropathy
Acronym: Assess CIPN
Status: Not yet recruiting | Type: Observational
Sponsor: Paracelsus Medical University (Other)
Collaborators: General Hospital Nuremberg & Paracelsus Medical University Nuremberg (Unknown)
Responsible Party: Principal Investigator, Florian Rieder, P.D.Dr. rer.nat., Paracelsus Medical University
Other Study IDs: UIPMR_CIPN
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN)
Keywords: CIPN, EORTC CIPN20, gait , balance, functional assessment, 9 hole peg test,
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CIPN patiients: CIPN
  Interventions: Diagnostic Test: Questionnaire and Physical Exam
- Healthy Controls: healthy
  Interventions: Diagnostic Test: Questionnaire and Physical Exam

INTERVENTIONS:
Diagnostic Test: Questionnaire and Physical Exam — Measurements: EORTC QLQ-CIPN 20 questionnaire, short physical performance test battery, gait and balance, 9 hole peg test, grip strength

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a severe side effect of several anti-cancer agents. Typical symptoms include tingling and hypoesthesia in the fingertips and/or toes, which substantially impair patients' quality of life and independence. Providing effective, evidence-based treatments for CIPN remains a major challenge in clinical practice. In a recent randomized clinical trial, our group demonstrated the effectiveness of electrotherapy in reducing both sensory and motor symptoms, as assessed by the EORTC-QLQ-CIPN20 questionnaire and CIPN grading according to CTCAE. However, these findings were based exclusively on patients' subjective self-reports (EORTC QLQ CIPN 20 and C-30). To more objectively evaluate treatment success, functional assessments that capture impairments in daily activities are needed.

In this cross-sectional comparison, we will conduct comprehensive functional assessments and correlate the results with patients' subjective ratings using the EORTC-QLQ-CIPN20, QLQ-C30, and CTCAE v5.0 grading. In addition, data from matched healthy controls will be collected and compared with those of CIPN patients. The findings of this study will contribute to the development of objective measures of functional limitations caused by CIPN and provide a valuable complement to patient-reported outcome obtained through validated questionnaires.

DETAILED DESCRIPTION:
Background Continuous advancements in diagnosis and treatment of cancer lead to rising numbers of cancer survivors and to increasing life expectancy (Jemal et al., 2023). However, the progress in systemic therapy also brings challenges in the management of side effects. Chemotherapy-induced peripheral neuropathy (CIPN) is one major complication of several anti-cancer therapies, especially of taxanes and platinum salts (Banach et al., 2017). In a meta-analysis of studies investigating taxanes and platinum salts, the average prevalence of CIPN was > 60% in the first 3 months after cessation of chemotherapy and about 30% after 6 months (Seretny et al., 2014). Symptoms usually begin during chemotherapy at a lower intensity and tend to increase if chemotherapy is continued. As a result, dose reductions and, ultimately, discontinuation of chemotherapy are frequently necessary in order to avoid high-grade CIPN, which hampers daily activities and diminishes quality of life (Bhatnagar et al., 2014). In most cases, initially only sensory function is affected (Kroigard et al., 2014), leading to symmetric tingling and hypoesthesia of fingertips and/or tiptoes. If the causing agent is continued, the CIPN symptoms could spread proximally to the fingers, hands, forearms and/or feet and legs, respectively. At a later stage, motor function is also affected, leading to a loss of strength and immobility (Kroigard et al., 2014). Within the first year after chemotherapy, symptoms may not resolve at all (Pachman et al., 2015) or may even intensify (Trivedi et al., 2023). The mechanisms leading to CIPN are complex, multifactorial and still not fully understood. The type of chemotherapeutic agent, its dose and treatment interval have all been shown to influence risk of CIPN (Was et al., 2022; Zajaczkowska et al., 2019). Microtubule disruption, oxidative stress and mitochondrial damage, altered ion channel activity, myelin sheath damage, DNA damage, immunological processes and neuroinflammation may play a key role (Was et al., 2022; Zajaczkowska et al., 2019). Unfortunately, there is still no effective pharmacological or non-pharmacological treatment of CIPN available. Several approaches with antidepressants, antiepileptics, magnesium, calcium, vitamins E and B6, glutamine, glutathione, N-acetyl-cysteine, omega-3 fatty acids, alpha lipoic acid, topical ketamine, acupuncture, or magnetic field therapy have not shown reproducible and significant relief of symptoms (Hershman et al., 2014; Hwang et al., 2020).

Recently, our group was funded by Paracelsus Medical University's Research Promotion Fund (PMU FFF) to investigate home-based electrotherapy using either transcutaneous electrical nerve stimulation (TENS) or high-tone external muscle stimulation (HTEMS) as a new strategy to improve CIPN symptoms (Schaffler-Schaden et al., 2020). This randomized clinical trial demonstrated a significant reduction in sensory and motor symptoms after eight weeks of home-based electrotherapy in both arms, measured with the EORTC QLQ-CIPN20 questionnaire and the grade of CIPN according to CTCAE v4.0 (Sassmann et al., 2024). Further, in secondary data analysis of this study (under review in Frontiers of Neurology), we observed that TENS and HTEMS improve CIPN symptoms differently. While TENS was effective in diminishing burning pain sensations, HTEMS was able to reduce numbness and tingling of feet and/or hands.

However, our data which indicated treatment success relies on patients' subjective ratings via specific questionnaires (e.g. EORTC QLQ CIPN 20 or C-30). These assessments are all well validated and reliable, but cannot objectively capture the restrictions on everyday life due to CIPN (Park et al, 2019). In order to assess objectively whether an intervention improves patients' everyday lives, additional assessments are needed. In the present study, a novel test battery using functional tasks will be developed and validated against in a cohort of CIPN patients and matched healthy controls. Once this test battery has been established, a prospective, interventional multicenter study is planned to examine the effects of electrotherapy.

Hereby, we hypothesize that (1) In CIPN patients, results of the functional tasks correlate to outcomes of the EORTC-QLQ-CIPN20 and EORTC-QLQ-C30 questionnaires.

(2) The performance of CIPN patients in the functional tasks will be lower compared to healthy controls.

Material and Methods Performance in selected functional tasks and subjectively rated functional impairments (EORTC-QLQ-CIPN20 and C30 questionnaires), will be assessed in patients undergoing chemotherapy as soon as CIPN-specific symptoms arise and in healthy matched controls. In a sub-group of the healthy controls, we will measure the functional tasks twice to assess the test-retest reliability.

The total duration of the study will be approximately 1 year. Subjects Inclusion criteria for CIPN patients

- Male and female patients with CIPN grade ≥ 2, according to Common Terminology Criteria for Adverse Events for peripheral sensory or motor neuropathy (CTCAE) version 5

- Age ≥ 18

- Ongoing or completed neuropathy-inducing chemotherapy

- Ability to stand and walk

- Ability to fill out a questionnaire Inclusion criteria for healthy controls

- Male and female adults (age ≥ 18)

- Ability to stand and walk

- Ability to fill out a questionnaire Exclusion criteria

- Pre-existing clinically manifest peripheral neuropathy prior to start of chemotherapy (e.g. caused by radiation or malignant plexopathy, lumbar or cervical radiculopathy, carpal tunnel syndrome, B12 deficiency, AIDS, monoclonal gammopathy, diabetes, heavy metal poisoning amyloidosis, syphilis, hyperthyroidism or hypothyroidism, inherited neuropathy, etc.)

- Acute or chronic injuries/ diseases of the musculoskeletal system affecting functional tests

- Acute or chronic cardiovascular diseases affecting functional tests

- Neurological disease affecting functional tests (for healthy controls)

- Neurological disease other than CIPN affecting functional tests (for CIPN patients) Recruitment PMU Salzburg CIPN Patients will be recruited and screened for eligibility at the Department of Internal Medicine III of the Paracelsus Medical University Salzburg. Careful review of inclusion and exclusion criteria, patient information and study enrollment will be done at the Institute of Physical Medicine and general Rehabilitation of the Paracelsus Medical University Salzburg. Healthy matched controls will be recruited among employees of the University Hospital Salzburg and the Paracelsus Medical University Salzburg (except employees of the Institute of Physical Medicine). Review of inclusion and exclusion criteria, participant information and study enrollment will be done at the Institute of Physical Medicine and general Rehabilitation of the Paracelsus Medical University Salzburg.

PMU Nuremberg CIPN patients will be recruited and screened for eligibility by physicians and study personnel of the Institute of Clinical Pharmacology, Paracelsus Medical University Nuremberg. Participants will include patients receiving chemotherapy with taxanes or platinum-agents at the Clinic of Gynecologic Oncology (Prof. Dr. C. Brucker), Clinic of Pneumology (Dr. M. Horneber), Clinic of Gastroenterology (Prof. Dr. M. Dechêne) and Clinic of Oncology (Prof. Dr. S. Knop). A careful review of inclusion and exclusion criteria, patient information and study enrollment will be provided by Clinical Pharmacology. Measurements can be performed at the premises of the Institute of Clinical Pharmacology on campus. Healthy matched controls will be recruited among employees of the Paracelsus Medical University and Klinikum Nuremberg.

Matching Healthy controls will be matched to CIPN patients according to following variables: sex, age, body mass, height, BMI, pre-illness activity level.

Measurements After inclusion CIPN patients and matched healthy controls will complete the EORTC-QLQ-CIPN20 and EORTC-QLQ-C30 questionnaires, the CIPN CTCAE grading as well as the functional tests at the Institute of Physical Medicine and general Rehabilitation of the PMU Salzburg or the Institute of Clincial Pharmacology in Nuremberg, respectively (figure 1). The measurements themselves will take approximately 90 minutes. A subsample of n=15 subjects of the matched healthy controls will perform the functional measurements twice to determine test-retest reliability.

Questionnaires The use of the CTCAE questionnaire is a standardized and validated tool to detect CIPN at an early stage (Le-Rademacher et al., 2017; Trotti et al., 2003). The combination with the EORTC QLQ-CIPN20 questionnaire is the best way to determine the clinical severity of the symptoms (Cavaletti et al., 2010). This questionnaire assesses impairments due to CIPN in the categories sensory function, motor functioning and autonomic function, is well standardized, objective, valid and reliable (Cavaletti et al., 2013). The EORTC QLQ-C30 questionnaire is designed for cancer patients and incorporates mainly five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting) and a global health status. This questionnaire has proven to be valid and reliable (Fayers P & Bottomley A, 2002).

Functional assessments Functional measurements contain gait and balance measurements, handgrip strength, the short physical performance test battery and the nine whole peg test. To measure gait and balance performance, patients wear pressure insoles (with 240 pressure sensors for each foot; Medilogic pressure insoles, Velamed/ Noraxon, Köln, Germany). Balance will be measured while patients are in a standing position on a flat surface and on a gymnastics mat for 30 seconds. Thereby, the movement of the center of pressure (COP) is measured. For the gait analysis, patients walk a distance of 5.5 m (distance of three gymnastics mats in a row) on a flat surface and on gymnastics mats with self-selected speed. Outcome parameters are step lengths, gait velocity, pressure distribution and COP movement. Reliability of the used measuring setup has been confirmed (Koch et al., 2016; Price et al., 2016). To test finger dexterity, patients will perform the nine whole peg test where nine small sticks have to be inserted into holes and pulled out again over time. This assessment is used for quantification of impaired upper extremity functions caused by various disorders (e.g. neurological disorders like multiple scleroses, post-stroke or polyneuropathy, (Feys et al., 2017; Johansson & Hager, 2019; Reddy et al., 2016). Handgrip strength is measured by pressing a handheld dynamometer to the maximum. This method is a valid tool to evaluate muscle strength of the upper extremities in healthy subjects and in various clinical conditions (Bobos et al., 2020) and correlates with CIPN symptom severity (Pattanshetty et al., 2020). The Short Physical Performance Test battery includes a balance test (standing in various positions for 10 seconds), a timed 4-meter walk test, and a timed chair rise test.

The following personal data will be additionally obtained: Age, sex, weight, height, smoking, consumption of alcohol, (former) profession, former and current physical activity, current ECOG status and medication.

Statistics Sample size was calculated using SPSS (IBM statistics) for Pearson-correlations. By assuming a power of 90% and a moderate correlation of 0.5 (Cohan´s d) as well as an alpha level of 95%, n = 37 patients are needed. Therefore, we plan to recruit n=20 CIPN patients in Salzburg and n= 20 CIPN patients in Nuremberg and the same number of healthy matched controls (20 at each location). Analyses will be elaborated in a prescribed statistical analysis plan. Normal distribution of data will be checked using the Shapiro-Wilk-Test. Group differences will be analyzed using t-tests for independent samples. Correlation analysis will be done by a person correlation or equivalent non-parametric procedures.Checks for linearity (which is expected regarding the variables) will be done optically by plotting the values in a scatter plot. If necessary, we will transform the data or use a spearman correlation model.The z transformation is also used to compare the performance of participants within the individual functional tests and to be able to perform factor analyses.

In addition, each individual functional variable will be examined for group differences between CIPN and healthy subjects. For this purpose, T-tests for independent samples will be used for normal distributions, otherwise adequate nonparametric methods will be used. To measure significant group differences, for a power of 0.80, an effect size d=0.6, and an alpha level of 5%, n= 37 individuals per group are needed (calculated in G*Power).

This cross-sectional comparison is of explorative nature and it is therefore not possible to determine primary and secondary endpoints a priori.

Randomization and Blinding Randomization into groups which receive additional tests or not will not be performed due to the exploratory design of this study. Blinding of patients is not possible, but investigators performing the functional test will not be given information about the medication, test results from questionnaires, or diagnoses. The inclusion of a control group will help to gauge the extent of the deficits.Expected Outcomes and Benefits Results of this pilot study will inform objective measurement of functional limitations due to CIPN and can supplement subjective ratings of patient reported outcomes. Thus, the effect of interventions on daily life functions can be evaluated in more detail. Our group is planning a multi-center study to investigate the effectiveness of electrotherapy for symptomatic treatment of CIPN. Adequately powered, the study will investigate operating areas (e.g. pain reduction vs mitigating tingling and numbness) of both electrical interventions, outcomes across different anti-cancer agents and reason for response or non-response to electrotherapy. Using the functional assessments tested in this present pilot study, we can investigate how improvements in CTCAE and EORTC-QLQ-CIPN20 / C30 scores translate to functional performance in daily life.

Patient Safety and Data Management In this cross-sectional comparison study the risk of potential harms for patients and healthy participants is very small. The functional tests will be supervised by experienced therapists and do not place any great strain on the cardiovascular or musculoskeletal systems. All tests, which are also performed on patients in routine clinical practice, will be performed at a University Hospital in Salzburg or Nuremberg and medical care is available on site if necessary. However, symptoms such as temporary exhaustion or muscle soreness may occur.

The balance measurements are performed between two support beams, which patients can hold onto if they loose balance. The gait measurements are supervised by a therapist who can intervene if necessary. These and similar measurements have been performed in our department for some time now, and there have been no incidents of patients falling. With these precautions in place, the risk of falling is extremely low, and insurance is therefore not necessary.

Translated with DeepL.com (free version) All obtained data will be pseudonymized (the coding list is stored electronically with restricted access to study personnel, only) and stored on secure hospital servers with access for study personal, only. An exchange of pseudonymized data between the study teams from Salzburg and Nuremberg will take place. The data will be processed and stored in accordance with the GDPR regulations.

Ethics The study will comply with the Declaration of Helsinki and will be designed according to the standards of good clinical practice. Approval of the study protocol / ICF will be obtained from the ethics committee of the state of Salzburg. Then, study documents will also submitted to the institutional review board at PMU in Nuremberg (Germany). Patient participation is voluntary and requires prior written informed consent. Before signing the consent form, each patient will be personally informed about the study objectives, procedures, potential risks and benefits, and data management. Patients may withdraw consent at any time without any disadvantage.

ELIGIBILITY:
Inclusion Criteria:

- Male and female patients with CIPN grade ≥ 2, according to Common Terminology Criteria for Adverse Events for peripheral sensory or motor neuropathy (CTCAE) version 5

- Age ≥ 18

- Ongoing or completed neuropathy-inducing chemotherapy

- Ability to stand and walk

- Ability to fill out a questionnaire Inclusion criteria for healthy controls

- Male and female adults (age ≥ 18)

- Ability to stand and walk

- Ability to fill out a questionnaire

Exclusion Criteria:

* Pre-existing clinically manifest peripheral neuropathy prior to start of chemotherapy (e.g. caused by radiation or malignant plexopathy, lumbar or cervical radiculopathy, carpal tunnel syndrome, B12 deficiency, AIDS, monoclonal gammopathy, diabetes, heavy metal poisoning amyloidosis, syphilis, hyperthyroidism or hypothyroidism, inherited neuropathy, etc.)

Acute or chronic injuries/ diseases of the musculoskeletal system affecting functional tests

- Acute or chronic cardiovascular diseases affecting functional tests

- Neurological disease affecting functional tests (for healthy controls)

- Neurological disease other than CIPN affecting functional tests (for CIPN patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CIPN patients from the paracleus medical university Healthy matched controls
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
correlation between questionnaire data abd functional assessments | 2 hours
  correlation between questionnaire data abd functional assessments
Correlations between questionnaire data and functional assessments | 2 hours

SECONDARY OUTCOMES:
Group differences in functional assessments between CIPN patients and helathy controls | 2 hours
  Group differences in functional assessments between CIPN patients and helathy controls

IPD SHARING:
Plan to Share IPD: No